CLINICAL TRIAL: NCT03183687
Title: Resident Wellness Initiative: Improving Physical Activity, Nutrition Education and Mental Health of Residents
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-1522
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2019-01

CONDITIONS: Mental Health Wellness 1
Keywords: neurosurgery; resident wellness; health; mental health; physical activity; physician health
MeSH Terms: conditions — Psychological Well-Being; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This wellness initiative is aimed to assess the activity level, sleep habits and nutrition status of resident physicians. The investigators will monitor for improvement in these areas with initiation of an exercise program suited to the lifestyle needs of resident physicians.

DETAILED DESCRIPTION:
The health and mental health benefits of physical activity, quality sleep and optimal nutritional habits are innumerable and widely reported. Unfortunately, resident physicians report participation in physical activity at reduced rates compared with the general population. Reasons for limited physical activity include fatigue and lack of free time to dedicate to exercise. The lack of exercise is combined with variable sleep patterns due to call schedules, as well as deterioration of nutritional habits, leads to weight gain and overall decline in the health of the resident physician population. Another neurosurgery department has implemented a similar program for their resident physicians and found improvements in weight, biometric markers and increased cardiovascular tolerance of physical activity.

The activity goals are derived from the 2013 the American Heart Association/American College of Cardiology Guidelines on lifestyle management to reduce cardiovascular risk, with considerations made for different levels of ability among the participants, as well as limitations time.

Fitness Protocol: The investigators will view any activity as better than no activity. The program will begin with activities geared toward the least fit/active resident to encourage participation from all levels of ability. The investigators will need options to increase intensity or difficulty for more advanced participants. Prior to introduction of the fitness regimen, the investigators would discuss appropriate progression of activity with a fitness expert. The proposed progression through various fitness goals is noted by type and timeline below.

Step Goal: Each participant will be asked to wear a fitness tracker to quantify steps walked per day, among other health parameters. Goals will be set for number of steps per day and per week, with incremental increase through the course of the program.

Cardiac Activity: Goals will be suggested for participants to complete cardiac activity through the course of their week. This may be running, which would overlap with the step goals, biking, or another cardiac exercise of the participants' preference. The goal will increase gradually over the course of the program.

Daily Challenge: A physical challenge will be extended to each participant to be completed every day, increasing in difficulty or repetitions through the month. This will be a simple task that could be performed without any equipment, such as (but not limited to) a plank hold, pushups or jumping jacks.

Weekly Workout: Workouts will be created by colleagues from appropriate departments (Kinesiology, Sports Performance) to be completed in a single ~30 minute setting or small 5-10 minute increments in order to be integrated into the physician lifestyle. These workouts will be completed on an individual basis and will be simple enough for completion in a small space, such as the call rooms, with access to hand weights, resistance bands and the stairwell.

Group Activities: Group activities will be planned once per month, with a focus on team building and physical activity. These group activities will be made available to non-study participants to encourage family attendance and participation in physical fitness. Some examples of proposed activities include soccer, sand volleyball, basketball.

Education: Colleagues from nutrition, neuropsychology and kinesiology will be invited for guest lectures on a monthly basis to improve resident education on topics such as making nutritionally smart choices and appropriate meal preparation, improving sleep hygiene, and how to incorporate activity into our currently lifestyles.

Study Timeline Pre-Program - distribution of surveys; biometric data obtained Month 1 - goal for steps. Group activity: movement safety. Month 2 - goal for steps + cardiac activity. Group activity. Month 3 - goal for steps + cardiac activity + daily challenge + improve sleep hygiene. Group activity. Repeat health surveys.

Month 4 - increase goal for steps + cardiac activity + daily challenge + weekly workout. Group activity.

Month 5 - goal for steps + cardiac activity + daily challenge + weekly workout + improve sleep habits. Group activity.

Month 6 - continuation of above goals + setting individual goals. Group activity.

Post-Program - distribution of surveys; biometric follow up data obtained.

ELIGIBILITY:
Current resident within the Neurosurgery Program in the Department of Neurological Surgery at the University of Wisconsin-Madison, provided they are willing to participate based on completion of informed consent.

Participants will likely be young adults in relatively good health status.

Inclusion criteria:

* resident within the Neurosurgery Program in the Department of Neurological Surgery at the University of Wisconsin-Madison
* ability to participate in light activity, and being willing to participate.

Exclusion criteria:

* Unable to participate in planned activities
* those not willing to participate
* non-resident department employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Current residents within the Neurosurgery Program in the Department of Neurological Surgery at the University of Wisconsin-Madison, provided they are willing to participate based on completion of informed consent. Participants will likely be young adults in relatively good health status. The study will be presented to the resident population as a group, as well as incoming residents in the future, with the hope that all are willing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the activity level of the resident physician population. | 3 years
  Resident physicians report participation in physical activity at reduced rates compared with the general population. Activity data will be obtained through the fitness tracker worn by each resident. The goal is to find improvements in weight (kg or Lb).

SECONDARY OUTCOMES:
Evaluate the mental health and sleep quality of the resident physician population. | 3 years
  Reasons for limited physical activity include fatigue and lack of free time to dedicate to exercise. The lack of exercise is combined with variable sleep patterns due to call schedules, leading to the overall decline in the health of the resident physician population. Sleep data will be obtained through the fitness tracker worn by each resident to monitor on a regular basis the sleep quality of the resident physician.
Monitor for improvement in basic health parameters with the implementation of a scheduled physical activity program and improved nutritional education | 3 years
  The activity goals are derived from the 2013 AHA/ACC Guidelines on lifestyle management to reduce cardiovascular risk, with considerations made for different levels of ability among the participants, as well as limitations of time.

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel P Brooks, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eckel RH, Jakicic JM, Ard JD, de Jesus JM, Houston Miller N, Hubbard VS, Lee IM, Lichtenstein AH, Loria CM, Millen BE, Nonas CA, Sacks FM, Smith SC Jr, Svetkey LP, Wadden TA, Yanovski SZ, Kendall KA, Morgan LC, Trisolini MG, Velasco G, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 AHA/ACC guideline on lifestyle management to reduce cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S76-99. doi: 10.1161/01.cir.0000437740.48606.d1. Epub 2013 Nov 12. No abstract available. PMID 24222015
- [Background] Fargen KM, Spiotta AM, Turner RD, Patel S. The Importance of Exercise in the Well-Rounded Physician: Dialogue for the Inclusion of a Physical Fitness Program in Neurosurgery Resident Training. World Neurosurg. 2016 Jun;90:380-384. doi: 10.1016/j.wneu.2016.03.024. Epub 2016 Mar 19. PMID 27001240
- [Background] Goetz K, Musselmann B, Szecsenyi J, Joos S. The influence of workload and health behavior on job satisfaction of general practitioners. Fam Med. 2013 Feb;45(2):95-101. PMID 23378076
- [Background] Lebensohn P, Dodds S, Benn R, Brooks AJ, Birch M, Cook P, Schneider C, Sroka S, Waxman D, Maizes V. Resident wellness behaviors: relationship to stress, depression, and burnout. Fam Med. 2013 Sep;45(8):541-9. PMID 24129866
- [Background] Levey RE. Sources of stress for residents and recommendations for programs to assist them. Acad Med. 2001 Feb;76(2):142-50. doi: 10.1097/00001888-200102000-00010. PMID 11158832
- [Background] Stanford FC, Durkin MW, Blair SN, Powell CK, Poston MB, Stallworth JR. Determining levels of physical activity in attending physicians, resident and fellow physicians and medical students in the USA. Br J Sports Med. 2012 Apr;46(5):360-4. doi: 10.1136/bjsports-2011-090299. Epub 2011 Dec 22. PMID 22194220
- [Background] Williams AS, Williams CD, Cronk NJ, Kruse RL, Ringdahl EN, Koopman RJ. Understanding the exercise habits of residents and attending physicians: a mixed methodology study. Fam Med. 2015 Feb;47(2):118-23. PMID 25646983